CLINICAL TRIAL: NCT05496075
Title: Observational Study on Clinical Efficacy and Safety of Orlistat in Reducing Uric Acid in Overweight/Obese Patients With Hyperuricemia
Brief Title: Orlistat Reduces Uric Acid in Overweight/Obese Patients With Hyperuricemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shanghai 10th People's Hospital (Other)
Responsible Party: Principal Investigator, Zhang Manna, Deputy Chief Physician, Shanghai 10th People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: orlistat reduces UA
Record Dates: First submitted 2022-08-08; First posted 2022-08-11 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Uric Acid
MeSH Terms: interventions — Orlistat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Orlistat group (Experimental): Orlistat was administered orally on the basis of lifestyle guidance.
  Interventions: Drug: Orlistat
- control group (Placebo Comparator): Orlistat placebo was administered orally on the basis of lifestyle guidance.
  Interventions: Drug: Orlistat placebo

INTERVENTIONS:
Drug: Orlistat — Orlistat was administered orally on the basis of lifestyle guidance . Orlistat: Take 0.12g (1 capsule) with or within one hour after meals, 3 times a day. Medication time course: continuous administration for a total of 12 weeks.
  Arms: Orlistat group
Drug: Orlistat placebo — Lifestyle guidance: low-purine diet; orlistat placebo: take 1 capsule with or within one hour after a meal, 3 times a day. Medication time course: continuous administration for a total of 12 weeks.
  Arms: control group

SUMMARY:
To clarify the uric acid-lowering efficacy of orlistat in overweight/obese patients with hyperuricemia, and to evaluate the safety of orlistat treatment

ELIGIBILITY:
Inclusion Criteria:

(Items 1, 2, and 4 meet at the same time, and items 3 and 5 meet one of them)

1. Obtain the informed consent of the subjects before any trial-related activities (including activities carried out to assess the eligibility of subjects);
2. Men or women over the age of 18 at the time of screening;
3. The diagnosis of hyperuricemia refers to the fasting of serum uric acid > 420umol/L (7 mg/dl) twice on different days under a normal purine diet.
4. The weight meets the following requirements (a or b): a) BMI ≥ 25.0 kg/m2; b) waist circumference, female ≥ 85 cm, male ≥ 90 cm.
5. Suffering from hyperuricemia and/or gout.-

Exclusion Criteria:

1. Use of drugs that may affect uric acid within 1 month before enrollment, including; benzbromarone, allopurinol, febuxostat, etc.;
2. Abnormal liver function, ALT and AST are more than 2.5 times the upper limit of normal;
3. Other diseases that affect glucose and lipid metabolism: hyperthyroidism, hypothyroidism, hypercortisolism, etc.;
4. Diabetic patients with poor blood sugar control: HbA1c>7%;
5. Chronic kidney disease or severe renal impairment, according to eGFR grading <45mL/min/1.73m2;
6. The life expectancy does not exceed 5 years;
7. Female subjects who are pregnant or plan to become pregnant within the next 24 weeks;
8. Those who are expected to be unable to complete the intervention follow-up in other circumstances;
9. If other drugs are used in combination, the drug dose should be kept stable for three months before enrollment;
10. Participated in other clinical trials within the past 4 weeks;
11. Use of drugs that affect body weight within 3 months before screening, including: systemic steroids (intravenous, oral or intra-articular), tricyclic antidepressants, psychiatric drugs or sedatives (eg, imipramine, amitriptyline, mirtazapine, paroxetine, phenelzine, chlorpromazine, thioridazine, clozapine, olanzapine, valproic acid, valproic acid derivatives, lithium salt), etc.;
12. Obesity caused by secondary diseases or drugs, including: elevated cortisol hormone (for example: Cushing's syndrome), obesity caused by pituitary and hypothalamus damage, obesity caused by reduction/discontinuation of weight loss drugs, etc.;
13. Inability to complete the exercise and for other reasons, the researcher believes that it is not suitable to participate in this researcher.-

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2022-08-26 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
level of uric acid | Month 3
  Change from Baseline Uric acid at 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Tenth People's hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Liu S, Lin X, Tao M, Chen Q, Sun H, Han Y, Yang S, Gao Y, Qu S, Chen H. Efficacy and safety of orlistat in male patients with overweight/obesity and hyperuricemia: results of a randomized, double-blind, placebo-controlled trial. Lipids Health Dis. 2024 Mar 11;23(1):77. doi: 10.1186/s12944-024-02047-7. PMID 38468241